CLINICAL TRIAL: NCT01487746
Title: Presence of Minor Anti Phospholipid Antibodies in Blood Samples of Ischemic Stroke Patients and Healthy Controls.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0125-11-MMC
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Ischemic Stroke
Keywords: APLA; APS; Stroke; minor anti body; major anti body; APLA antibodies in Serum
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples of Stroke patients withdrawned within 36 hrs since stroke evoked. Healthy controls
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- treatment: Stroke patients
- Controls: healthy controls

SUMMARY:
The investigators expect to find higher levels of both classical and minor antiphospholipid (APL) antibodies among the stroke cases. Furthermore, the investigators expect to find not only classical APLA but also minor antibodies.

The investigators believe that minor antibodies have a major role in the hypercoagulability state.

ELIGIBILITY:
Inclusion Criteria:

* stroke diagnosis
* blood sampling within 36hrs from the event
* written agreement

Exclusion Criteria:

* a stroke, MI or major operation prior to the current stroke
* hypercoagulable state known in this patient
* a severe chronic disease known at the time of the stroke
* an infection on arrival (based on anamnesis, physical exam and lab tests)
* thrombolytic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: on a bank of 207 stroke patients serum samples, and also on 40 healthy controls. The samples were collected during the acute phase of the ischemic event.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir health center, Kfar Saba, Israel